CLINICAL TRIAL: NCT03079089
Title: Sequential Chemotherapy Prior Conditioning Reduced Intensity: Study Routine Care in Haploidentical Allogeneic Hematopoietic Stem Cells in Patients With Relapsed or Refractory Lymphoid Hematological Disorders
Brief Title: Sequential Conditioning in Haploidentical Transplantation for Hematopoietic Stem Cells in Patients With Relapsed or Refractory Lymphoid Hematological Disorders
Acronym: LY-SET-HAPLO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Association for Training, Education, and Research in Hematology, Immunology, and Transplantation (Other)
Responsible Party: Principal Investigator, Pr Mohamad MOHTY, Principal investigator, Association for Training, Education, and Research in Hematology, Immunology, and Transplantation
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2016-A00861-50
Record Dates: First submitted 2017-02-16; First posted 2017-03-14 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Refractory or Relapsed Lymphoid Haemopathy
Keywords: Allogenic cell stem transplant; Sequential chemotherapy; Haploidentical transplant

STUDY DESIGN:
Intervention Model Description: Patients with refractory or relaps lymphoid hematological disorders
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Relapsed or refractory lymphoid hematological disorders (Other): Patients in refractory or relapses with an indication of allo-HSC used the combination of an SET followed by the RIC with the PDLI
  Interventions: Drug: Sequential Packaging (SET); Drug: Transfusion graft; Drug: Prevention of GVHD; Drug: Care supports; Drug: Lymphocyte injection of prophylactic donor (PDLI)

INTERVENTIONS:
Drug: Sequential Packaging (SET) — Sequential chemotherapy: - Thiotepa 5 mg/kg/day for 1 day (D-13) -Cyclophosphamide 400 mg/m²/day for 4 days (J-12 to J-9)- Etoposide 100 mg/m²/day for 4 days (J-12 to J-9) Repos days J-8 and J-6 Reduced-intensity conditioning (RIC)-Fludarabine 30 mg/m²/day for 5 days (J-5 to D-1)- Busulfan IV 3.2 mg/kg/day for 2 days (J-5 and J-4)- Anti-lymphocyte serum (Thymoglobuline) 2.5 mg / kg / day for 2 days (J-3 and J-2)
Drug: Transfusion graft — Graft of peripheral stem cells is preferred at DO
Drug: Prevention of GVHD — * Cyclophosphamide 50mg/ kg/day on days D + 3 and D + 5 - Cyclosporine A (CSA; 3 mg / kg / day IV from D+6)
  * Mycophenolate mofetil (MMF; 30 mg/kg/ day, maximum x2 1g / day from day J+6)
Drug: Care supports — According to the protocols of each center
Drug: Lymphocyte injection of prophylactic donor (PDLI) — According to the protocols of each center. In the absence of clinical indication against-disease (GVHD), phasing MMF between days D + 35 and D + 56, then phasing APF between D + 62 and D + 90
  - PDLI: 3 injections from the D + 120 patients who discontinued immunosuppressive therapy for ≥ 1 month and having no active GVHD or history of acute GVHD grade> II.

SUMMARY:
Allogeneic hematopoietic stem cell transplantation (allo-HSCT) is the only treatment option with a significant chance of healing in lymphoid hematological refractory or multiple relapses after chemotherapy. However, all patients with an indication of allo-HSC can not benefit because of two limitations: the toxicity of the treatment and graft shortage available.

For patients refractory or in relapses with an indication of allo-HSC, used the combinaison of an SET followed by the reduced-intensity allo-HSC (RIC) has shown some interesting results.

A post-transplant immune modulation with prophylactic injections of donor lymphocytes (PDLI) showed its effectiveness to decrease the risk of relapse while having a lower toxicity than chemotherapy

ELIGIBILITY:
Inclusion Criteria:

* Patients with an indication of allo-HSC for a lymphoid hematological malignancy like Hodgkin's lymphoma, non hodgkin's lymphoma b cell (mantle follicular, diffuse large cells, marginal zone,MALT) or T (peripheral T whithout specificity, anaplasic, angio-immunoblastic, natural killer cells, gamma / delta T cells, Sezary's syndrome, primitive cutaneous T), prolymphocytic leukemia, chronic lymphocytic leukemia, waldenström's disease and for which a therapeutic strategie combining a sequential chemotherapy followed by the reduced-intensity conditioning(SET RIC + PDLI) is decided
* Patients at least in partial response (standard criteria) after a rescue treatment the day of evaluation at 1 month before the conditioning
* Advanced age ≥ 18 to <60 years
* Cardiac ejection fraction of the left ventricle ≥ 45%
* Lung function - free diffusion capacity for carbon monoxide ≥ 50% of predicted value
* Creatinine clearance ≥ 50 ml / min depending on the CKD-EPI formula
* Availability of an HLA haploidentical donor in the family
* Collection of non-opposition

Exclusion Criteria:

* Invasion of uncontrolled CNS
* Availability of an HLA identical family donor who agreed to donate hematopoietic stem cells OR non-related donor HLA-compatible 10/10 on HLA-A alleles, B, C, and DRB1 DQB1 available and ready to give in 4 weeks to make a decision allograft
* Presence in the patient HLA-specific antibodies directed against an antigen HLA haploidentical donor family
* Karnofsky score <70%
* Patient HIV positive
* Hepatitis B or C or chronic active
* Uncontrolled infection at the time of start packing
* Contraindication to the use of treatments provided by the protocol
* Previous history of allo-HSC
* No beneficiary of a social security scheme.
* life expentancy estimated less than 1 month by investigator

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2017-06-30 (Actual); Primary Completion 2023-09-11 (Actual); Study Completion 2023-09-11 (Actual)

PRIMARY OUTCOMES:
Overall survival (OS) | 2 years after transplantation
  Describe efficacy and safety of the combination of an SET followed by the RIC with post-transplant immune modulation by PDLI in patients with refractory or relaps lymphoid hematological refractory or multiple relapses lymphoid hematological disorders

SECONDARY OUTCOMES:
Partial or complete remission rate by standard criteria relapse incidence and death related to the disease and free survival | 90 days and then 6, 12 and 24 months after transplantation
  Describe the efficacy of this therapeutic strategy in terms of remission of disease, incidence of relapse and relapse-free survival
Cumulative incidence of death not related to relapse | 90 days and then 12 and 24 months after transplantation
  Describe not related to relapse mortality
Cumulative incidence of acute and chronic graft against host disease (GVHD) | 100 days and then 12 and 24 months after transplantation
  Describe the incidence of acute and chronic graft against host disease (GVHD)
Number of patients for whom PDLI was possible and number PDLI / patient ; incidence, severity and treatment of possible secondary GVHD in these patients | 2 years after transplantation
  Describe the feasibility of prophylactic injections of donor lymphocytes (PDLI)
Immune reconstitution post-transplantation in the peripheral blood | 30, 90 and 180 days after transplantation
  Immune reconstitution will be determined by CD4 lymphocyte, CD8, T regulators, Natural Killer cells and B cells levels in the peripheral blood
Tolerance of this therapeutic strategy | 90 days and the 6, 12 and 24 month after transplantation
  The tolerance will be evaluated by:
  1. The cumulative incidence of death not related to relapse at 90 days, 1 year and 2 years after transplantation
  2. The cumulative incidence of acute and chronic graft against host disease (GVHD)
  3. The incidence of advert events

CONTACTS AND LOCATIONS:
Locations (1):
- Service d'hématologie clinique Hôpital Saint Antoine, Paris, France

IPD SHARING:
Plan to Share IPD: No